CLINICAL TRIAL: NCT01602536
Title: Twitter-enabled Mobile Messaging for Smoking Relapse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cornelia Pechmann, Principal Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20107990; 1R34DA030538-01A1 (NIH)
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Smoking
Keywords: twitter; quit smoking; smoking cessation; social media; peer support
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Twitter (Experimental): Experimental participants are assigned a 20-person twitter quit-smoking group to interact with, are instructed to use Twitter-enabled interactive peer messaging,and are sent daily messages to encourage interaction. The baseline intervention 'smoking cessation aides' is also provided.
  Interventions: Behavioral: smoking cessation aides; Behavioral: Twitter
- Control (Active Comparator): Control participants are not assigned to a twitter group. The baseline intervention 'smoking cessation aides' is also provided.
  Interventions: Behavioral: smoking cessation aides

INTERVENTIONS:
Behavioral: smoking cessation aides — All participants will receive 8 weeks of free nicotine patches, referral to the NCI's online Smokefree.gov Quit Guide, and instruction to set a quit date within 8 days of study start.
Behavioral: Twitter — Twitter quit-smoking group
  Arms: Twitter

SUMMARY:
We conducted a two-arm (test vs. control, N=160) randomized controlled trial of small, private, online support groups for quitting smoking with 20 people per group who were seeking to quit smoking. A novel feature was a bot (auto-messenger) that posted a daily cessation-related discussion topic in each group, timed to the group's quit date.

DETAILED DESCRIPTION:
Smoking relapse rates remain high, innovative strategies are needed to lower them, and web-based social networking may help like Twitter. This developmental research examined whether providing virtual (web-based) social support to smokers, through Twitter-enabled interactive peer texting, could help smokers quit and avoid relapses. Twitter is a free social networking and micro-blogging service, one of the most advanced and novel technologies available today that can provide social support to smokers, and it provides free texting to groups. It is global and has many features that are associated with treatment success including interactive, multi-way, live messaging and mobile accessibility, because the messages go instantly to mobile phones and to the web. It can provide an innovative way to reach smokers who might otherwise not seek treatment, and it can be extended to other health domains. From June 2012 through 2014, we conducted a two-condition randomized controlled trial. All participants in this trial (N=160) received 8 weeks of free nicotine patches, referral to the NCI's online Smokefree.gov Quit Guide, and instruction to set a quit date within 1 week of study start. Participants were also randomly assigned at the individual level to one of two conditions: (1) a virtual or online quit-smoking group on Twitter where the group members were instructed to use interactive peer messaging to help them quit and stay quit, or (2) a control group condition where the group members were not given this instruction or a Twitter group. In total, there were 4 Twitter groups and 4 control groups with 20 smokers randomly assigned to each group (i.e., N=80 test, N=80 control). In the Twitter groups, a bot (auto-messenger) posted a daily cessation-related discussion topic in each group, timed to the group's quit date. The primary outcome was self-reported 7-day point prevalence abstinence that was sustained at 7, 30 and 60 days after the quit date. Participants' posts, their virtual and face-to-face social networks, and several other possible mediating and moderating variables were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* must have smoked 100 cigarettes during their lifetime
* must currently smoke 5 or more cigarettes a day
* must be in the preparation stage of quitting smoking
* ages 18-59 years
* English speaking
* have a mobile phone with an unlimited texting plan and internet access
* use text messaging at least once a week
* use Facebook daily
* have an active email account
* live in the continental USA

Exclusion Criteria:

* a medical condition that is contra-indicated for nicotine replacement therapy:
* pregnant
* breast feeding
* a recent heart attack
* an irregular heartbeat
* high blood pressure not controlled with medication
* skin allergies to adhesive tape or serious skin problems
* taking a prescription medicine for depression or anxiety
* use drugs or marijuana regularly
* live in the same household with another participant

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Pechmann, PhD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Hosted Study Website Tweet2Quit@Merage.Uci.Edu, Irvine, California
  - University of California Irvine, Irvine, California

REFERENCES:
- [Derived] Pechmann C, Delucchi K, Lakon CM, Prochaska JJ. Randomised controlled trial evaluation of Tweet2Quit: a social network quit-smoking intervention. Tob Control. 2017 Mar;26(2):188-194. doi: 10.1136/tobaccocontrol-2015-052768. Epub 2016 Feb 29. PMID 26928205
- [Derived] Pechmann C, Pan L, Delucchi K, Lakon CM, Prochaska JJ. Development of a Twitter-based intervention for smoking cessation that encourages high-quality social media interactions via automessages. J Med Internet Res. 2015 Feb 23;17(2):e50. doi: 10.2196/jmir.3772. PMID 25707037
- See also: tweet2quit website — http://tweet2quit.merage.uci.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Twitter | Control
Started | 80 | 80
Completed | 65 | 70
Not Completed | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twitter | Control | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 35.35 (10.55) | 36.00 (9.16) | 35.68 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 61 | 116
  Male | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 7-day Point Prevalence Abstinence From Smoking That Was Sustained at 60 Days After the Quit Date
Description: self-reported 7-day point prevalence abstinence from smoking that was sustained at 60 days after the quit date, based on survey
Time Frame: 60 days after quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Twitter | Control
Number analyzed (Participants) | 65 | 70
Participants | 26 | 14

2. Secondary Outcome: Level of Engagement Based on Tweet Volume
Description: level of engagement based on tweet volume which is observed in support groups
Time Frame: 100 days total
Population: all participants were observed to assess their tweeting (posting) behavior
Measure: Mean (Standard Deviation); unit: social media posts
Arm/Group | Twitter | Control
Number analyzed (Participants) | 80 | 80
social media posts | 58.86 (68.02) | 0 (0)

ADVERSE EVENTS:
Time Frame: 3 MO.
Arm/Group | Twitter | Control
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes